CLINICAL TRIAL: NCT01223066
Title: A Multi-center, Non-interventional, Prospective Study to Monitor Long Term Safety in Female Subjects After Treatment With Macrolane Volume Restoration Factor 20 and/or Macrolane Volume Restoration Factor 30 in the Breasts.
Brief Title: Macrolane Prospective Survey
Status: Withdrawn | Type: Observational
Why Stopped: no patients recruited
Sponsor: Galderma R&D (Industry)
Collaborators: Pharma Consulting Group AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 31GB0906
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2012-11

CONDITIONS: Females Recently Treated With Macrolane VRF in the Breasts
Keywords: Macrolane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women treated with Macrolane in the breasts

SUMMARY:
The study objective is to evaluate the long term safety when Macrolane Volume Restoration Factor is used in female breasts in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Females recently treated with Macrolane Volume Restoration Factor in the breasts.
* Signed informed consent

Exclusion Criteria:

* There are no exclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participating clinics will ask women who have been treated with Macrolane in the breasts in clinical practice, to participate in this survey.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedén, Md PhD, Principal Investigator — Akademikliniken Stockholm
Locations (1):
- Akademikliniken, Stockholm, Sweden